CLINICAL TRIAL: NCT05451199
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Single and Multiple AscendingDose Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ICP-488 in Healthy Subjects and Patients With Psoriasis
Brief Title: A Clinical Study of ICP-488 in Healthy Subjects and Patients With Psoriasis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICP-CL-01001
Record Dates: First submitted 2022-06-24; First posted 2022-07-11 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICP-488 (Experimental): Single ascending doses of ICP-488 tablet; Multiple ascending doses of ICP-488 tablet; Part3 Patients with Psoriasis:ICP-488 tablet.
  Interventions: Drug: ICP-488
- Placebo (Placebo Comparator): Single ascending doses of placebo; Multiple ascending doses of placebo; Part3 Patients with Psoriasis of placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ICP-488 — ICP-488 will be administered as tablet
  Arms: ICP-488
Drug: Placebo — Matching placebo will be administered as tablet
  Arms: Placebo

SUMMARY:
This is a Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Single and Multiple AscendingDose Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ICP-488 in Healthy Subjects and Patients With Psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed informed consent, and was able to communicate well with the investigator and can complete the study according to the study requirement.
2. Body mass index (BMI) between 18-26 kg/m2, the weight of male subject should not be less than 50 kg, and the weight of female subject should not be less than 45 kg.
3. The results of laboratory tests during the screening period are within the normal reference values of the population or study site;Or the results were slightly off but within acceptable limits, and the investigator evaluated that they were not clinically significant.
4. Fertility status: Female subjects who are infertile (i.e. physically unable to conceive, including postmenopausal or surgically infertile women);Male subjects and their partners must agree to use effective contraception for the entire study period and for 28 days after the last medication or for five half-lives, and male subjects shall not donate sperm during this period.
5. Male or female subjects aged ≥ 18 years and ≤ 65 years；
6. Diagnosis of plaque psoriasis；
7. All of the following 3 criteria are met at screening and randomization:

1）Psoriasis Area and Severity Index (PASI) ≥ 12; 2）Physician Global Assessment (PGA) ≥ 3; 3）Body surface area (BSA) affected by psoriasis ≥ 10%.

8. The subject is a candidate to receive systemic therapy and/or phototherapy.

Exclusion Criteria:

1. Unable to follow the study protocol requirements.
2. Evidence or history of clinically significant disease, or evidence or history of allergic disease.
3. Subjects with clinically significant gastrointestinal dysfunction that may affect drug intake, transport or absorption.
4. Acute disease state within 14 days before administration.
5. Currently or within 6 months prior to administration experiencing a severe infection or having a long-term or recurrent infection disease
6. Subjects and/or first-degree relatives have a genetic immune deficiency.
7. Major trauma or surgery within 3 months prior to the first administration.
8. Previous medical history of tuberculosis; The presence of investigator-judged signs or symptoms of active tuberculosis and the chest imaging showed active pulmonary tuberculosis at screening ；T-spoT test (T-SPOT) was positive at screening.
9. Urine drug test positive.
10. Alcoholic
11. Subjects who have used tobacco/cigarettes or tobacco/cigarette products within 3 months prior to the first administration.
12. Subjects who donated more than 500 ml of blood (excluding plasma) within 56 days before the first dose, or planned to donate blood or blood components during the study period or within 1 month after the study finished.
13. Use of any other study drug specified in the protocol within 30 days prior to initial administration or within 5 half-lives(refer to whichever is longer).
14. Any traditional Chinese medicine (TCM) and over-the-counter (OTC) drugs, vitamins, systemic steroid hormone therapy, immunosuppressant or modulator therapy, hormone replacement therapy, and other food supplements or herbs were used 30 days before the first dose until follow-up visit.
15. Consume any food or drink containing caffeine within 48 hours prior your first administration.
16. Last use of stron , moderate and weak CYP1A2/CYP3A4 inhibitors or inducers less than 5 half-lives before the first dose of study drug, or planning to take medications, dietary supplements, or foods
17. Diet or dietary treatment within 30 days prior to initial administration or have significant change in eating habits.
18. Eat smoked charcoal fire foods (such as Carbon barbecue,etc) within 1 week prior to the study.
19. Any positive showed in the lab result of syphilis specific antibody, hepatitis C antibody (HCV-Ab), hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb) or human immunodeficiency virus serological antibody (HIV-Ab) during screening.
20. Received vaccination with live virus vaccine, live attenuated vaccine or any live virus component is administered within 6 weeks prior to initial administration, or during the planned study period or within 8 weeks after the end of the study.
21. Non-plaque forms of psoriasis.
22. Drug-induced psoriasis.
23. Are taking or require oral or injectable corticosteroids for any medical condition.
24. Clinically significant test results at the time of screening that, in the investigator's judgment, may cause unacceptable risk to the participant.
25. History of active tuberculosis，active hepatitis B virus、active hepatitis C virus or Syphilis infection.
26. Clinically severe, progressive, or uncontrolled disease at screening； Pregnant female subjects.
27. breastfeeding female subjects.
28. Other situations judged by the investigator to be unsuitable to join this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events during treatment, and withdrawal from treatment due to adverse events | Single ascending dose: 1day；Multiple ascending dose: 28 days

SECONDARY OUTCOMES:
Cmax | Single ascending dose: 1day；Multiple ascending dose: 28 days
Psoriasis Area and Severity Index （PASI） | Day1,Day7,Day14,Day21,Day28,Day35,Day42,Day56
Body Surface Area （BSA） | Day1,Day7,Day14,Day21,Day28,Day35,Day42,Day56
Static Physician's Global Assessment （sPGA） | Day1,Day7,Day14,Day21,Day28,Day35,Day42,Day56
Peak Pruritus Numerical Rating Scale （PP-NRS） | Day1-Day14, Day21, Day28, Day35, Day42, Day56
Dermatology quality of life index （DLQI） | Day1,Day7,Day14,Day21,Day28,Day35,Day42,Day56

CONTACTS AND LOCATIONS:
Overall Officials: Qianjin Lu, Principal Investigator — Hospital for Skin Diseases, Chinese Academy of medical Sciences
Locations (7):
- China (7):
  - The Second Hospital of Anhui Meidcal University, Hefei, Anhui
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Nanyang First People's Hospital, Nanyang, Henan
  - Shiyan Renmin Hospital, Shiyan, Hubei
  - Hospital for Skin Diseases, Institute of Dermatology, Chinese Academy of medical Sciences, Peking Union Medical College, Nanjing, Jiangsu
  - Yanbian University Hospital, Yanji, Jilin
  - Hangzhou First People's Hospital, Hangzhou, Zheajing